CLINICAL TRIAL: NCT03318640
Title: Effect of Mindfulness (MBSR) on the Parasympathetic System and Cognition in Schizophrenia
Brief Title: Mindfulness and Cognition in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low inclusion rates
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1708181; 2017-A02921-52 (Other: ANSM)
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Schizophrenia
Keywords: schizophrenia; mindfulness; parasympathetic system
MeSH Terms: conditions — Schizophrenia | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Comparison between treated group or not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Patient will have 8 sessions (1h30) of mindfulness based on Kabat-Zinn program during one month.
  Interventions: Behavioral: Mindfulness
- Control (No Intervention): Patient will have usual medical care.

INTERVENTIONS:
Behavioral: Mindfulness — Patient will have 8 sessions (1h30) of mindfulness based on Kabat-Zinn program during one month
  Arms: Mindfulness

SUMMARY:
Mindfulness (innovative and integrative practice in care) allows the individual to adapt his/her behavior (physical and emotional), in a stressful environment, by regulating cardiac activity, especially the parasympathetic system. In schizophrenia, despite the positive effect of treatments on symptoms (delusions and hallucinations), patients have altered markers of the parasympathetic (high frequency, HF) system. The investigator propose a session of Mindfulness Based Stress Reduction (MBSR) for patients suffering from schizophrenia in order to measure the impact on the parasympathetic system (HF), self-awareness (being well in one's body and being aware of their own actions; EASE) and cognition (attention) in relation to the management of conflicts or emotions. The study compare with patients who receive a session of techniques based on the management of emotions and social cognition (cinemotion, Michael's Game and Tom Remed).

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia (men only)
* aged 18-55
* with no change in antipsychotic medication and clinical status within four weeks prior to the study
* affiliates or entitled to a social security scheme
* who have given their informed consent before participating in the study.

Exclusion Criteria:

* History of head trauma, neurological disease or not stabilized serious physical illness
* Disorders related to the use of a psychoactive substance, as defined by the DSM-IV (abuse, dependence or withdrawal) within 6 months
* Beta blocking and anti-arrhythmic medications.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
High Frequency spectral power | 2 months
  High Frequency spectral power

SECONDARY OUTCOMES:
Score | 2 months
  Score of PANSS (POSITIVE AND NEGATIVE SYNDROME SCALE)
Score | 2 months
  The five facet questionnaire Mindfulness Questionary Freiburg

CONTACTS AND LOCATIONS:
Overall Officials: Anne GROSSELIN, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No